CLINICAL TRIAL: NCT02517320
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of MT-3995 in Patients With Diabetic Nephropathy
Brief Title: Efficacy and Safety of MT-3995 in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-3995-J05
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MT-3995 Low (Experimental)
  Interventions: Drug: MT-3995 Low
- MT-3995 Middle (Experimental)
  Interventions: Drug: MT-3995 Middle
- MT-3995 High (Experimental)
  Interventions: Drug: MT-3995 High
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-3995 Low
  Arms: MT-3995 Low
Drug: MT-3995 Middle
  Arms: MT-3995 Middle
Drug: MT-3995 High
  Arms: MT-3995 High
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of MT-3995 in subjects with diabetic nephropathy, compared with placebo, using urine albumin- to-creatinine ratio (UACR) in the first morning void urine sample as an indicator.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Glycated hemoglobin(HbA1c) values (National Glycohemoglobin Standardization Program : NGSP) ≤10.5%
* estimated glomerular filtration rate(eGFR) of ≥30 mL/min/1.73 m2
* The median UACR of the first morning void urine samples is ≥50 mg/g Cr and <300 mg/g Cr
* Stable blood pressure(diastolic blood pressure (DBP) <100 mmHg and stable systolic blood pressure (SBP) <160 mmHg)

Exclusion Criteria:

* Type 1 diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes.
* A diagnosis of non-diabetic renal disease.
* A following serum potassium level.

  * eGFR of 30-59mL/min/1.73m2; serum potassium level of <3.5 or >4.7 mmol/L,
  * eGFR of ≥60mL/min/1.73m2: serum potassium level of <3.5 or >5.0 mmol/L
* symptomatic and clinically significant hypotension(diastolic blood pressure(DBP)<50mmHg and systolic blood pressure(SBP)<110mmHg)
* QT prolongation or torsades de pointes, or, a history or family history of QT prolongation or torsades de pointes
* New York Heart Association (NYHA) Class III or IV heart failure

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change form baseline in UACR | Week 24

SECONDARY OUTCOMES:
Change in UACR classification | From baseline to 24 weeks
Change in renal function | From baseline to 24 weeks
Change in serum potassium | From baseline to 24 weeks
Adverse events | From baseline to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Hokkaido, Japan

REFERENCES:
- [Derived] Wada T, Inagaki M, Yoshinari T, Terata R, Totsuka N, Gotou M, Hashimoto G. Apararenone in patients with diabetic nephropathy: results of a randomized, double-blind, placebo-controlled phase 2 dose-response study and open-label extension study. Clin Exp Nephrol. 2021 Feb;25(2):120-130. doi: 10.1007/s10157-020-01963-z. Epub 2020 Sep 24. PMID 32974732